CLINICAL TRIAL: NCT01523834
Title: A Phase II Study of Oral Panobinostat in Adult Patients With Diffuse Large B-cell Lymphoma Relapsed/Refractory After High-dose Chemotherapy With Autologous Stem Cell Transfusion (ASCT) or Not Eligible for ASCT
Brief Title: Oral Panobinostat Adult Patients DLBCL Relapsed/Refractory Stem Cell Transfusion (ASCT) or Not Eligible for ASCT
Acronym: FIL_PanAL10
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_PanAL10; 2011-000175-13 (EudraCT Number)
Record Dates: First submitted 2011-06-22; First posted 2012-02-01 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Diffuse Large B-cell Lymphoma (DLBCL); Panobinostat; Patients with relapsed/refractory DLBCL.
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Panobinosat (Experimental): The treatment is divided in three phases: induction phase (course 1 to 6), consolidation phase (courses 7 to 12), maintenance phase (from course 13 until the end of therapy for any reason). The duration of a treatment course will be 28 days. The first dose of panobinostat in course 1 defines day 1 of the treatment cycle, and each cycle thereafter will begin 28 days later.
  Treatment:
  Panobinostat should be taken p.o. at the dose of 40 mg/day three-times every week (QW) (e.g., on Monday, Wednesday, and Friday or Tuesday, Thursday, and Saturday), as part of a 4 week (28 days) treatment cycle.
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat — Induction Phase: Patients will receive panobinostat for 6 courses (1 course = 28 days). Consolidation phase (courses 7-12). Maintenance phase (course 13-end of therapy).
  Panobinostat should be taken p.o. at the dose of 40 mg/day 3-times every week (QW) as part of a 4 week treatment cycle. The dose of panobinostat may be modified: the 1st dose adjustment consists in the modification of drug administration from 3 times every week (QW) to 3 times every other week (QOW). Levels lower than 30 mg 3 times QOW is not permitted.
  Other Names: LBH589

SUMMARY:
Treatment of adult patients with Diffuse Large B-cell Lymphoma (DLBCL), relapsed or refractory to previous CHOP-R (or CHOP-R like regimen) front line therapy, relapsed or refractory to second or subsequent salvage therapies which included high dose therapy with autologous stem cell support (ASCT).

Treatment of adult patients with DLBCL relapsed or refractory to front line therapy with CHOP-R (or CHOP-R like regimen) or subsequent treatments, who are not consider eligible for ASCT consolidation because of age, co-morbidities, impossibility to perform ASCT.

The trial is conducted according to the optimal two-stage design of Simon with alpha 0.05 and beta 0.10, considering the following two hypotheses: first a response rate (RR) less than 10% is of no further interest; and second, an RR 30% is clinically meaningful. In the initial stage, 18 patients have to enter onto the study. If less than 3 responses (</=2 in 18) will be observed, the trial would be terminated. Otherwise, accrual will continue to a total of a maximum of 35 patients. At the end of the trial, if 6 or fewer responses will occur among the 35 patients (</= 6 in 35), it will be concluded that the regimen is not worthy of further investigations for that group of patients.

The treatment is divided in three phases: induction phase (course 1 to 6), consolidation phase (courses 7 to 12), maintenance phase (from course 13 until the end of therapy for any reason).

DETAILED DESCRIPTION:
Overview Of Study Design This is a prospective, multicenter phase II trial designed to evaluate the safety and activity of the panobinostat in patients with relapsed/refractory diffuse large B-cell lymphoma (DLBCL). Study design The trial is conducted according to the optimal two-stage design of Simon with alpha 0.05 and beta 0.10, considering the following two hypotheses: first a response rate (RR) less than 10% is of no further interest; and second, an RR 30% is clinically meaningful. In the initial stage, 18 patients have to enter onto the study. If less than 3 responses (£ 2 in 18) will be observed, the trial would be terminated. Otherwise, accrual will continue to a total of a maximum of 35 patients. At the end of the trial, if 6 or fewer responses will occur among the 35 patients (£ 6 in 35), it will be concluded that the regimen is not worthy of further investigations for that group of patients. The treatment is divided in three phases: induction phase (course 1 to 6), consolidation phase (courses 7 to 12), maintenance phase (from course 13 until the end of therapy for any reason). Study duration This study is expected to start in February 2011. The last patient is expected to be enrolled at the end of January 2013. Considering a possible treatment duration of 24 months, this trial is due to be completed by January 2015.

Objectives:

Primary objective 1. To explore the antitumor activity of panobinostat in term of overall response (OR) at the end of the induction phase (i.e. month 6 from the beginning of panobinostat) Secondary objectives

1. To explore the antitumor activity of panobinostat in terms of Complete Response (CR)
2. To assess the time to response (TTR)
3. To evaluate Progression Free Survival (PFS)
4. To assess the safety and tolerability of panobinostat
5. To evaluate the Overall Survival (OS) Exploratory objectives

1. To study the impact of pharmacogenetics in predicting the response to panobinostat 2. To study the impact of immunohistochemical patterns and patient's specific gene expression and response to panobinostat 3. To assess the correlation between "telomeric asset" and response to panobinostat

ELIGIBILITY:
Inclusion Criteria:

1. Patient age is ≥ 18 years
2. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
3. Patient has a history of DLBCL according to the WHO classification
4. Patient has progressive disease after receiving at least CHOP-R or CHOP-R like first line regimen, standard second line therapy (DHAP, ESHAP, ICE or similar salvage regimens) inclusive ASCT
5. Patient has progressive disease after receiving at least CHOP-R or CHOP-R like first line regimen and is not considered eligible for intensive salvage therapy including ASCT because of age, co-morbidities, impossibility to perform ASCT
6. Patient undergoes at baseline new lymphnode or other pathologic tissue biopsy for confirmation of diagnosis and biologic studies; bone marrow biopsy is not adequate for this purpose and should be performed only for staging. Patients with primary refractoriness, not eligible for intensive salvage therapy including ASCT, who performed a previous biopsy with stored frozen material 6 months or less before enrolment into the study do not have to repeat a new biopsy
7. Patient has at least one site of measurable nodal disease at baseline ≥ 2.0 cm in the longest transverse diameter as determined by CT scan (MRI is allowed only if CT scan can not be performed). Note: Patients with bone marrow involvement are eligible, but this criteria alone should not be used for disease measurement
8. Patient has the following laboratory values (labs may be repeated, if needed, to obtain acceptable values before screen fail):

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L [SI units 1.5 x 109/L]
   * Platelet count ≥ 100 x 109/L
   * Serum potassium, magnesium, phosphorus, sodium, total calcium (corrected for serum albumin) or ionized calcium within normal limits (WNL) for the institution
   * Serum creatinine ≤ 1.5 x ULN
   * Serum bilirubin ≤ 1.5 x ULN (or ≤ 3.0 x ULN, if patient has Gilbert syndrome)
   * AST/SGOT and/or ALT/SGPT ≤ 2.5 x upper limit of normal (ULN) or ≤ 5.0 x ULN if the transaminase elevation is due to disease involvement
9. Clinically euthyroid. Note: Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism
10. Written informed consent was obtained from the patient prior to any study-specific screening procedures
11. Patient has the ability to swallow capsules or tablets
12. Practice acceptable birth control.

Exclusion Criteria:

1. Patient has a history of prior treatment with a DAC inhibitors including panobinostat
2. Patient will need valproic acid for any medical condition during the study or within 5 days prior to the first panobinostat treatment
3. Patient has been treated with monoclonal antibody therapy (e.g., rituximab or anti CD-30 antibody, etc.) within 4 weeks of start of study treatment
4. Patient has been treated with any other anti lymphoma therapy within 3 weeks of start of study treatment
5. Patient is using any anti-cancer therapy concomitantly
6. Patient has been treated with > 5 prior systemic lines of treatment
7. Patient has received prior radiation therapy ≤ 4 weeks or limited field radiotherapy ≤ 2 weeks prior to start of study treatment
8. Patient treated with allogeneic hematopoietic stem cell transplant with active progressive cGVHD; patient has received DLI ≤ 6 weeks prior to start of study treatment; patient is planned to receive DLI
9. Patient has a history of another malignancy ≤ 3 years before study entry, with the exception of non-melanoma skin cancer and carcinoma in situ of uterine cervix
10. Patient has a history of CNS involvement with lymphoma
11. Patient has impaired cardiac function including any of the following:

    * Complete left bundle branch block or use of a permanent cardiac pacemaker, congenital long QT syndrome, history or presence of ventricular tachyarrhythmias, clinically significant resting bradycardia (<50 beats per minute), QTcF > 450 msec on screening ECG, or right bundle branch block + left anterior hemiblock (bifascicular block)
    * Presence of unstable atrial fibrillation (ventricular heart rate >100 bpm). Patients with stable atrial fibrillation are allowed in the study provided they do not meet the other cardiac exclusion criteria
    * Previous history angina pectoris or acute MI within 6 months
    * Congestive heart failure (New York Heart Association functional classification III-IV)
12. Patient has any other clinically significant heart disease (e.g., uncontrolled hypertension)
13. Patient has an impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of panobinostat (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, obstruction, or stomach and/or small bowel resection)
14. Patient has unresolved diarrhoea ≥ grade 2
15. Patient has any other concurrent severe and/or uncontrolled medical condition(s) (e.g., uncontrolled diabetes mellitus, active or uncontrolled infection, chronic obstructive or chronic restrictive pulmonary disease including dyspnoea at rest from any cause) that could cause unacceptable safety risks or compromise compliance with the protocol
16. Patient has a known history of HIV seropositivity
17. Patient has active HBV hepatitis. The following categories of patients HBV positive but with non evidence of active hepatitis may be considered for the study and treated with panobinostat (see also Section 8.12 of the study protocol):

    * patient is HBsAg + with HBV DNA < 2000 UI/ml (inactive carriers); HBV DNA > 2000 UI/ml is criteria of exclusion
    * patient is HBsAg - HBsAb +
    * patient is HBsAg - but HBcAb +
18. Patients with HCV active hepatitis are excluded from the study. Patient with no evidence of active hepatitis and/or advanced chronic liver disease according to liver biopsy or fibro-scan evaluation may be included into the study (see also Section 8.12 of the study protocol)
19. Patient is using medications that have a relative risk of prolonging the QT interval or of inducing "Torsade de Pointes", where such treatment cannot be discontinued or switched to a different medication prior to starting study drug
20. Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not willing to use a double method of contraception during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months or had menses any time in the preceding 12 consecutive months. WOCBP must have a negative serum pregnancy test at baseline
21. Male patient whose sexual partner(s) are WOCBP who are not willing to use a double method of contraception, one of which includes a condom, during the study and for 3 months after the end of treatment
22. Patient does not have before entering into the study a new lymphnode or other pathologic tissue biopsy for confirmation of diagnosis and biologic studies; bone marrow biopsy is not adequate for this purpose and should be performed only for staging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Levis, MD, Principal Investigator — Fondazione Italiana Linfomi - ETS
Locations (10):
- Italy (10):
  - Azienda Ospedaliera SS. Antonio e Biagio e C. Arrigo, Alessandria
  - Istituto di Ematologia ed Oncologia Medica A. Seragnoli Policlinico S. Orsola, Bologna
  - Spedali Civili, Brescia
  - Ematologia I, A.O.U. San Martino, Genova
  - Ospedale Umberto I - DH Oncoematologico, Nocera Inferiore
  - Divisione di Ematologia Università Avogadro, Novara
  - AO Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - A.O. Città della Salute e della Scienza (Ematologia Univ), Torino
  - A.O. Città della salute e della scienza (S.C. Ematologia), Torino
  - AO Universitaria di Udine, Udine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first enrolment: 14th June 2011 Date of last completed: 3rd April 2017
  All patients (35) were enrolled in Italy.
Groups:
- Panobinosat: The treatment is divided in three phases: induction phase (course 1 to 6), consolidation phase (courses 7 to 12), maintenance phase (from course 13 until the end of therapy for any reason). The duration of a treatment course will be 28 days. The first dose of panobinostat in course 1 defines day 1 of the treatment cycle, and each cycle thereafter will begin 28 days later.
  Treatment:Panobinostat should be taken p.o. at the dose of 40 mg/day three-times every week (QW) (e.g., on Monday, Wednesday, and Friday or Tuesday, Thursday, and Saturday), as part of a 4 week (28 days) treatment cycle.
  Panobinostat: Induction Phase: Patients will receive panobinostat for 6 courses (1 course = 28 days). Consolidation phase (courses 7-12). Maintenance phase (course 13-end of therapy).
  Panobinostat should be taken p.o. at the dose of 40 mg/day 3-times every week (QW) as part of a 4 week treatment cycle. The dose of panobinostat may be modified: the 1st dose adjustment consists in the modificatio
Period: Overall Study
Arm/Group | Panobinosat
Started | 35 (Started Induction Phase)
Consolidation Phase | 7 (Started Consolidation Phase)
Maintenance Phase | 6 (Started Maintenance Phase)
Completed | 4
Not Completed | 31

BASELINE CHARACTERISTICS:
Population: Adult patients with diffuse large B-cell lymphoma relapsed/refractory after high-dose chemotherapy with autologous stem cell transfusion (ASCT) or not eligible for ASCT.
Groups:
- Panobinosat: The treatment is divided in three phases: induction phase (course 1 to 6), consolidation phase (courses 7 to 12), maintenance phase (from course 13 until the end of therapy for any reason). The duration of a treatment course will be 28 days. The first dose of panobinostat in course 1 defines day 1 of the treatment cycle, and each cycle thereafter will begin 28 days later.
  Treatment: Panobinostat should be taken p.o. at the dose of 40 mg/day three-times every week (QW), as part of a 4 week (28 days) treatment cycle. Panobinostat: Induction Phase: Patients will receive panobinostat for 6 courses (1 course = 28 days). Consolidation phase (courses 7-12). Maintenance phase (course 13-end of therapy). Panobinostat should be taken p.o. at the dose of 40 mg/day 3-times every week (QW) as part of a 4 week treatment cycle.
Arm/Group | Panobinosat
Number analyzed (Participants) | 35
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73 [65 to 75.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 21
Region of Enrollment [Number; unit: participants]
  Italy | 35

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) at the End of the Induction Phase
Description: ORR is defined as the proportion of patients achieving a Complete Response (CR) or Partial Response (PR) according to the Cheson 1999 response criteria
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Panobinosat: The treatment is divided in three phases: induction phase (course 1 to 6), consolidation phase (courses 7 to 12), maintenance phase (from course 13 until the end of therapy for any reason). The duration of a treatment course will be 28 days. The first dose of panobinostat in course 1 defines day 1 of the treatment cycle, and each cycle thereafter will begin 28 days later.
  Treatment: Panobinostat should be taken p.o. at the dose of 40 mg/day three-times every week (QW) (e.g., on Monday, Wednesday, and Friday or Tuesday, Thursday, and Saturday), as part of a 4 week (28 days) treatment cycle
  Panobinostat: Induction Phase: Patients will receive panobinostat for 6 courses (1 course = 28 days). Consolidation phase (courses 7-12). Maintenance phase (course 13-end of therapy).
  Panobinostat should be taken p.o. at the dose of 40 mg/day 3-times every week (QW) as part of a 4 week treatment cycle. The dose of panobinostat may be modified: the 1st dose adjustment consists in the modificatio
Arm/Group | Panobinosat
Number analyzed (Participants) | 35
percentage of participants | 17.1 [6.6 to 33.6]

2. Secondary Outcome: Complete Response (CR) Rate
Description: Proportion of CR at the end of the induction phase according to the Cheson 1999 response criteria
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Panobinosat: The treatment is divided in three phases: induction phase (course 1 to 6), consolidation phase (courses 7 to 12), maintenance phase (from course 13 until the end of therapy for any reason). The duration of a treatment course will be 28 days. The first dose of panobinostat in course 1 defines day 1 of the treatment cycle, and each cycle thereafter will begin 28 days later.
  Treatment:
  Panobinostat: Induction Phase: Patients will receive panobinostat for 6 courses (1 course = 28 days). Consolidation phase (courses 7-12). Maintenance phase (course 13-end of therapy).
  Panobinostat should be taken p.o. at the dose of 40 mg/day 3-times every week (QW) as part of a 4 week treatment cycle. The dose of panobinostat may be modified: the 1st dose adjustment consists in the modification of drug administration from 3 times every week (QW) to 3 times every other week (QOW). Levels lower than 30 mg 3 times QOW is not permitted.
Arm/Group | Panobinosat
Number analyzed (Participants) | 35
percentage of participants | 11.4 [3.2 to 26.7]

3. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as the time from enrolment to Overall Response
Time Frame: 36 months
Population: as for baseline characteristics
Measure: Median (Full Range); unit: months
Arm/Group | Panobinosat
Number analyzed (Participants) | 9
months | 2.6 [1.8 to 12.0]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from enrolment to disease progression or relapse or death from any cause
Time Frame: 36 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panobinosat
Number analyzed (Participants) | 35
months | 2.4 [1.4 to 7.0]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from enrolment to death from any case
Time Frame: 36 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panobinosat
Number analyzed (Participants) | 35
months | 7.6 [3.0 to 12.7]

ADVERSE EVENTS:
Time Frame: 6 years
Description: We used the Common Terminology Criteria for Adverse Events v. 4.0 (CTCAE) for the coding of adverse events.
Arm/Group | Panobinosat
All-Cause Mortality (participants affected / at risk) | 29/35
Serious Adverse Events (participants affected / at risk) | 12/35
Other Adverse Events (participants affected / at risk) | 8/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panobinosat (N=35)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Acute renal injury (Renal and urinary disorders) | 1 (1) — Pancytopenia and Gastroenteritis with dehydratation and acute renal failure.
Parossistic atrial fibrillation and congestive heart failure (Cardiac disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Nodular lesion rigth breast
Chest Pain (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Subocclusive syndrome (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Nausea, vomit, diarrea, ipoK+, atc prolonged (Metabolism and nutrition disorders) | 1 (1)
Paralysis of arms (Nervous system disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panobinosat (N=35)
Disease progression (General disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No